CLINICAL TRIAL: NCT03550625
Title: Computer Assisted Selection of Serrated Adenomas and Neoplastic Polyps - a New Clinical Draft
Acronym: CASSANDRA I
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: CASSANDRA I
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Polyps; Adenoma Colon; Automatic Judgement; Colonic Neoplasms
MeSH Terms: conditions — Polyps; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Colonic polyps
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Routine Colonoscopy Cohort: Photographies of polyps for creation of computer program
  Interventions: Diagnostic Test: Computer program

INTERVENTIONS:
Diagnostic Test: Computer program — No study specific intervention. Still images of polyps are collected. Histopathological reports of the resected polyps will be evaluated in order to create a computer program.

SUMMARY:
The aim of the study is to develop a computer program which is able to classify different entities of colorectal polyps on the basis of optical polyp features. In the end, the computer program shall differentiate between (i) hypeplastic polyps, (ii) adenomas and (iii) serrated adenomas .

In the first phase of the study a computer program will be established which aims to distinguish between the above mentions entities on the basis of optical features derived from still images. A machine learning apporach will be used for creating the program. Afterwards, in a second phase of the study, still images of 100 polyps (not used in the first phase) will be presented to the computer program. Quality of the computer program will be tested by calculating the accuracy for differentiating the three different polyp types. The gold standard for true polyp diagnoses will be based on histopathological diagnoses of the polyps. The same pictures of 100 polyps will also be presented to human experts. Experts will also predict histopathological diagnoses on the basis of optical polyps featurs. Accuracy of computer-decisions and human expert predictions will be compared. The establishment of a well- functioning computer program is the primary aim of the study.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* patients >= 18 years

Exclusion Criteria:

* pregnant women
* indication for colonoscopy: inflammatory bowel disease
* indication for colonoscopy: polyposis syndrome
* indication for colonoscopy: emergency colonoscopy e.g. acute bleeding
* contraindication for polyp resection e.g. patients on warfarin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for routine colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the computer- made optical diagnosis of each colorectal polyp | participants data will be followed for the duration of creating the computer program (an expected average of 2 month)
  The predicted polyp histology (made optically by the computer program) will be assessed; the predicted diagnosis will be compared with the histopathological diagnosis (gold standard) after resection of the polyp;

IPD SHARING:
Plan to Share IPD: No